CLINICAL TRIAL: NCT04883008
Title: A Multicenter Post-Market Study for the Evaluation of the CorPath® GRX technIQ Automated Movements in Percutaneous Coronary Interventions
Brief Title: NAVIGATE GRX Study
Status: Terminated | Type: Observational
Why Stopped: Sponsor business decision and low enrollment
Sponsor: Corindus Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 104-09466
Record Dates: First submitted 2021-04-13; First posted 2021-05-12 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Intervention: CorPath GRX with technIQ automated movements enabled (technIQ ON)
  Interventions: Device: CorPath GRX with technIQ automated movements enabled (technIQ ON)
- Control: CorPath GRX with technIQ automated movements disabled (technIQ OFF).
  Interventions: Device: CorPath GRX with technIQ automated movements disabled (technIQ OFF).

INTERVENTIONS:
Device: CorPath GRX with technIQ automated movements enabled (technIQ ON) — The CorPath GRX System is intended for use in the remote delivery and manipulation of guidewires and rapid exchange catheters, and remote manipulation of guide catheters during percutaneous coronary and vascular procedures.
  TechnIQ automated movements are software-based automation of common maneuvers that interventionalists perform when manipulating catheters, guidewires, and devices by hand. In this group, automated movements will be enabled and used at the discretion of the interventionalist.
  Groups: Intervention
Device: CorPath GRX with technIQ automated movements disabled (technIQ OFF). — The CorPath GRX System is intended for use in the remote delivery and manipulation of guidewires and rapid exchange catheters, and remote manipulation of guide catheters during percutaneous coronary and vascular procedures.
  TechnIQ automated movements are software-based automation of common maneuvers that interventionalists perform when manipulating catheters, guidewires, and devices by hand. In this group, automated movements will be disabled.
  Groups: Control

SUMMARY:
The objective of the present study is to detail the results of robotic-assisted PCI using technIQ automated movements in real-world clinical practice.

DETAILED DESCRIPTION:
This multi-center, international, randomized, open-label, post-market study will enroll subjects to detail the results of robotic-assisted PCI using technIQ automated movements in real-world clinical practice by randomized comparison with a cohort of subjects undergoing robotic-assisted PCI with technIQ automated movements disabled. A secondary objective is to describe the learning curve associated with using technIQ.

ELIGIBILITY:
Inclusion Criteria:

* Male or nonpregnant female aged ≥ 20 years.
* Patients with coronary artery disease with clinical indication for Percutaneous Coronary Intervention (PCI).
* The subject has been informed of the nature of the study, agrees to its provisions and has provided written informed consent.

Exclusion Criteria:

* Failure/inability/unwillingness to provide informed consent.
* In the opinion of the investigator, the subject is deemed unsuitable for robotic PCI due to clinical status or anatomic characteristics.
* Acute STEMI within 72 hours pre-procedure.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The targeted population is subjects with coronary artery disease and with a clinical indication for PCI.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-02-07 (Actual)

PRIMARY OUTCOMES:
Major Clinical and Angiographic Complications (MCAC) | 72 hours post-procedure or until immediately prior to discharge from the index procedure hospitalization, whichever occurs first.
  The rate of the combined MCAC endpoint (a composite of MACE and Major Clinical and Angiographic Complications) in the technIQ ON group is not significantly higher than in the technIQ OFF group.
Technical Success | During the Procedure
  Residual stenosis of <30% in all target lesions with final TIMI (Thrombolysis In Myocardial Infarction) flow grade 3 by angiographic core lab analysis, AND absence of unplanned manual conversion.

SECONDARY OUTCOMES:
PCI procedure time | During the Procedure
  Time between insertion of guide catheter and final removal of guide catheter.
Procedure success | 72 hours post-procedure or until immediately prior to discharge from the index procedure hospitalization, whichever occurs first.
  The rate of procedure success in the technIQ ON group is not significantly lower than that in the technIQ OFF group.
Major adverse cardiovascular events (MACE), | 72 hours post-procedure or until immediately prior to discharge from the index procedure hospitalization, whichever occurs first.
  Reported as a composite and components of Cardiac Death, Target Vessel MI, and Target Vessel Revascularization (TVR).
Major angiographic complications | During the Procedure
  Reported as perforation(Type 1, 2, 3) or flow-limiting dissection (Type E, F).
Serious Adverse Events (SAE) | Procedure through 72 hours postprocedure or hospital discharge (whichever occurs)
  All Serious Adverse Events (SAEs) from the start of the CorPath GRX PCI procedure through 72 hours postprocedure or hospital discharge (whichever occurs) first will be summarized
Guidewire Wiring Time | During the Procedure
  The time required to advance the guidewire from the tip of the guide catheter to the final target distal to the lesion.
Fluoroscopy Time to Cross Lesion | During the Procedure
  The fluoroscopy time required to advance the guidewire from the tip of the guide catheter to the final target distal to the lesion.
Contrast Used to Cross Lesion | During the Procedure
  The amount of contrast (in ml) required to advance the guidewire from the tip of the guide catheter to the final target distal to the lesion.
Total Procedural Time | During the Procedure
  The time from the start of the sheath insertion to complete removal of the final guide catheter.
Total Fluoroscopy Time | During the Procedure
  The total fluoroscopy time during the procedure as recorded by an Imaging System.
Subject Radiation Exposure | During the Procedure
  Dose-area-product (DAP) as recorded during the procedure
Subject Radiation Dose | During the Procedure
  air kerma (AK) as recorded during the procedure.
Contrast Fluid Volume | During the Procedure
  The total contrast volume used during the procedure.
Planned Manual Conversion (PMC) | During the Procedure
  Planned manual conversion (PMC) is disengagement of the robotic drive to use bedside manipulation of either the guide catheter, guidewire, or delivery system that was prespecified in the procedural plan (e.g., to accommodate adjunctive devices or procedural techniques that are not compatible with the robotic platform, such as intravascular ultrasound or atherectomy devices). This will be assessed by a questionnaire.
Unplanned Manual Conversion (UMC) | During the Procedure
  Unplanned manual conversion (UMC) is disengagement of the robotic drive to use bedside manipulation of either the guide catheter, guidewire, or delivery system that was not prespecified in the procedural plan, and that was due to inability to navigate to the target lesion as intended, cross the target lesion as intended, treat the target lesion as intended, retract the CorPath GRX system as intended, or other CorPath system device malfunction; or any clinical condition that requires rapid medical intervention. This will be assessed by a questionnaire.
Partial Manual Assistance (PMA) | During the Procedure
  Partial manual assistance (PMA) is the use of manual techniques that were not prespecified in the procedural plan and do not meet the definition of unplanned manual conversion (e.g., unplanned use of manual techniques to accommodate adjunctive devices or procedural techniques that are not compatible with the robotic platform). These will be assessed by a questionnaire.
Device Malfunction | During the Procedure
  The device malfunction will report the inadequacy of the medical device with respect to its identity, quality, durability, reliability, usability, safety, or performance. Investigators are instructed to report all device deficiencies and device malfunctions using the device malfunction form in the EDC.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Fajadet, MD, Principal Investigator — Groupe Cardiovasculaire Interventionnel, Clinique Pasteur
Locations (1):
- Intercard Sp. Z o.o., Nowy Sącz, Poland

IPD SHARING:
Plan to Share IPD: No